CLINICAL TRIAL: NCT06187831
Title: Changes in Central Venous Catheterization Bleeding Events After Implementing a Lower Trigger For Platelet Transfusion - an Observational Study
Brief Title: Bleeding Events Before vs After Lowering Departmental Platelet Transfusion Trigger
Acronym: OBS-PLATE
Status: Recruiting | Type: Observational
Sponsor: Thomas Kander (Other)
Responsible Party: Sponsor-Investigator, Thomas Kander, Associate Professor, Region Skane
Organization: Region Skane (Other)
Other Study IDs: OBS-PLATE
Record Dates: First submitted 2023-12-17; First posted 2024-01-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Bleeding; Central Line Complication; Thrombocytopenia; Hematologic Diseases
MeSH Terms: conditions — Hemorrhage; Thrombocytopenia; Hematologic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Before the change of the departmental pre-procedural platelet transfusion trigger for CVC placement: Patients ≥18 years of age admitted to a hematological ward at the current department, with an indication for CVC placement will be eligible for inclusion in the study
- After the change of the departmental pre-procedural platelet transfusion trigger for CVC placement: Patients ≥18 years of age admitted to a hematological ward at the current department, with an indication for CVC placement will be eligible for inclusion in the study

SUMMARY:
Central venous catheters are essential when administering treatment for hematological conditions. Many patients have a decreased platelet count which increases the risk for bleeding complications.

Baarle et al. recently published a randomized controlled study where withholding prophylactic platelet transfusions before CVC placement in patients with a platelet count of 10,000 to 50,000 per cubic millimeter did not meet the predefined margin for non-inferiority for postprocedural bleeding events (PMID: 37224197). However, bleedings grade 2 (defined as bleeding that requires external compression) were included despite lacking clinical significance.

The aim of the present study is to investigate whether lowering the preprocedural platelet transfusion trigger from 50x10^9/L to 10x10^9/L for insertions of central venous catheters remains safe with regards to postprocedural bleeding events of grade 3-4.

DETAILED DESCRIPTION:
This is a single-center, retrospective, observational study. All adult hematologic patients receiving a central venous catheter in the department of intensive and perioperative care at Skåne University Hospital in Lund, Sweden will be eligible for inclusion.

Current Swedish guidelines recommend a pre-procedural platelet transfusion trigger of 50x10^9/L to decrease the risk of bleeding during and after the procedure. However, these guidelines are based on data from an era when the landmark technique was predominant, and the bleeding complication incidence has decreased with the widespread use of real-time ultrasound guidance. Thus, our departmental pre-procedural platelet transfusion trigger for CVC placement was lowered from 50 to 10x10^9/L in March 2023. This corresponds to the threshold commonly used in hematologic patients to prevent spontaneous bleeding.

This study is set to investigate if the incidence of grade 3-4 postprocedural bleeding events have increased after the change in platelet transfusion trigger from 50x10^9/L to 10x10^9/L before the insertion of a CVC in hematologic patients.

Approximately 110 CVCs are placed annually in hematological patients at the current institution. Retrospective data will be extracted from the electronic charts and prospective data will be collected continuously. Intervention checkpoints will be put in place to control for grade 3-4 bleeding events:

1. The transfusion trigger will remain at 10x10^9/L provided that the incidence of post-procedural grade 3-4 bleeding events in patients with a pre-procedural platelet count of 10-49 x10^9 is less than three in six months, less than four in one year or less than five in two years.
2. The transfusion trigger will be increased to 30x10^9/L if the incidence of post-procedural grade 3-4 bleeding events in patients with a pre-procedural platelet count of 10-49 x10^9 is more than two in six months, more than three in one year or more than four in two years.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Indication for central venous catheter placement.
* Patients admitted to a hematological ward at the current department

Exclusion Criteria:

* Death within 24h after insertion of CVC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients ≥18 years of age admitted to a hematological ward at the current department, with an indication for CVC placement, will be eligible for inclusion in the study.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-02-26 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-04-20 (Estimated)

PRIMARY OUTCOMES:
Incidence of bleeding events grade 3 and 4 | Up to 24 hours after insertion of a central venous catheter
  Incidence of bleeding events grade 3 and 4 according to the National Cancer Institute Common Terminology criteria for Adverse events (CTCAE), version 5.0.

SECONDARY OUTCOMES:
Incidence of bleeding events grade 2 | Up to 24 hours after insertion of a central venous catheter
  Incidence of bleeding events grade 2 according to the National Cancer Institute Common Terminology criteria for Adverse events (CTCAE), version 5.0
Number of patients receiving pre-procedural platelet transfusion Number of patients receiving pre-procedural platelet transfusion | From 24 hours before to 24 hours after insertion of a central venous catheter
  Number of patients receiving pre-procedural platelet transfusion
Number of preprocedural units of platelet transfusions | From 24 hours before to 24 hours after insertion of a central venous catheter
  Number of preprocedural units of platelet transfusions

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Kander, PhD, Principal Investigator — Region Skåne Sweden
Locations (1):
- Thomas Kander, Lund, Lunds Universitet, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Upon reasonable request, de-identified individual participant data from this clinical trial will be shared to facilitate scientific collaboration.
Supporting Information: Study Protocol, CSR
Time Frame: After the publication of the study up to 3 years after the publication of the study
Access Criteria: Researchers may submit requests through the specified channel, detailing the purpose and proposed analyses. Approved applicants will sign a data access agreement, ensuring responsible and transparent use of the data.